CLINICAL TRIAL: NCT00277875
Title: The Effect of Vascular Distensibility on Endothelial-Dependent Vasoreactivity in Patients With Systolic Hypertension Before and After Receiving Oral Alagebrium for 8 Weeks.
Brief Title: STRETCH Study: Effect of Distensibility on Endothelial-Dependent Vasoreactivity in Patients With ISH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Synvista Therapeutics, Inc (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: ALT-711-0217
Record Dates: First submitted 2006-01-13; First posted 2006-01-18 (Estimated); Last update posted 2009-08-27 (Estimated); Status verified 2006-01

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular; Flow-Mediated Vasodilation (FMD); Pulse Perfusion-Mediated Vasodilation (PPMV); Endothelial Function; Heart Failure; Local Distensibility; Arterial Stiffening; Augmentation Index (AI); Aging; Isolated Systolic Hypertension; Advanced Glycation Endproducts; Vascular Stiffness
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure; Isolated Systolic Hypertension | interventions — alagebrium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ALT-711 (alagebrium chloride)

SUMMARY:
Determine whether increasing arterial distensibility by decreasing advanced glycation end-product (AGE) cross-link components of vascular stiffness improves (a) endothelial-mediated vasoreactivity at rest, as assessed by flow-mediated vasodilation (FMD), and (b) endothelial-mediated vasoreactivity after exercise, as assessed by pulse perfusion-mediated vasodilation (PPMV).

DETAILED DESCRIPTION:
* Explore several independent variables as potential independent predictors of vascular stiffness and endothelial function. These parameters include patient age, body mass index, gender, renal disease, history of cardiovascular disease, serum cholesterol, and antihypertensive medication use.
* Provide insight into nitric oxide-dependent endothelial function in the setting of increased arterial stiffness by determination of substances in the nitric oxide signaling pathway (specifically, levels of serum cGMP; serum nitrate and nitrite; and serum asymmetric dimethylarginine [ADMA], an endogenous inhibitor of nitric oxide synthase).
* Provide insight into changes in AGE levels and collagen metabolism in response to alagebrium therapy [specifically, AGEs: pentosidine, carboxymethyllysine, carboxyethyllysine, furosine; Collagen markers: procollagen I carboxyterminal propeptide (PICP), procollagen type I N terminal propeptide (PINP), cross-linked carboxyterminal telopeptide of Type I collagen (ICTP), n-terminal propeptide of type III procollagen (PIIINP)].
* Provide insight into changes in markers of inflammation in response to alagebrium therapy [specifically, free and total serum matrix metalloproteinase-1(MMP-1), free tissue inhibitor of metalloproteinase 1 (TIMP1), intercellular adhesion molecule-1 (ICAM), P-selectin, von Willebrand factor (vWf), interleukin-6 (IL-6), and high-sensitivity C reactive protein (hs CRP)].

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 50 years of age or greater.
2. Diagnosed with systolic hypertension (systolic blood pressure >140 mm Hg and (less than or equal to) 200 mm Hg, and a diastolic blood pressure (less than or equal to) 95 mm Hg) and elevated pulse pressure (systolic blood pressure [SBP] minus diastolic blood pressure [DBP] greater than 60 mm Hg).
3. Normal left ventricular function (ejection fraction >55%) at baseline (Visit 3).
4. Able to perform bicycle exercise.
5. Able to read, understand and sign the informed consent after the nature of the study has been explained.
6. If sexually active, the patient agrees to use reliable contraception while participating in this study. If a woman, is surgically sterilized or post-menopausal, or has a negative serum pregnancy test.

Exclusion Criteria:

1. Aortic stenosis, prior known coronary artery disease (including myocardial infarction), cerebrovascular accident, or peripheral vascular disease.
2. Uncontrolled hypertension (SBP > 200/ DBP > 95 mm Hg).
3. Atrial fibrillation, diabetes mellitus treated with insulin, or chronic lung disease.
4. Any additional condition(s) which, in the opinion of the investigator, would prohibit the patient from completing the study, or not be in the best interest of the patient.
5. Treatment with nitrates, or a change in antihypertensive medications within the last 1 month.
6. Treatment with any investigational drug within 1 month prior to study drug administration.
7. Previous exposure to alagebrium.
8. AST (SGOT) or ALT (SGPT) > 2x normal limit.
9. Serum creatinine > 2.0 ng/mL.
10. Cigar/cigarette smoking.
11. Necessity to use smokeless tobacco or nicotine-containing products, or to consume caffeine, alcohol, or antioxidants starting at midnight prior to study clinic visits. NOTE: Water is allowed ad libitim.
12. Positive drug screen.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2004-02; Primary Completion 2004-12 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Endothelial function
Local distensibility
Arterial stiffening
Augmentation index (AI)
Markers of endothelial function, vascular inflammation and collagen synthesis.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Zieman, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Background] Kass DA, Shapiro EP, Kawaguchi M, Capriotti AR, Scuteri A, deGroof RC, Lakatta EG. Improved arterial compliance by a novel advanced glycation end-product crosslink breaker. Circulation. 2001 Sep 25;104(13):1464-70. doi: 10.1161/hc3801.097806. PMID 11571237
- [Background] Liu ZR, Ting CT, Zhu SX, Yin FC. Aortic compliance in human hypertension. Hypertension. 1989 Aug;14(2):129-36. doi: 10.1161/01.hyp.14.2.129. PMID 2759675
- [Background] Corretti MC, Anderson TJ, Benjamin EJ, Celermajer D, Charbonneau F, Creager MA, Deanfield J, Drexler H, Gerhard-Herman M, Herrington D, Vallance P, Vita J, Vogel R; International Brachial Artery Reactivity Task Force. Guidelines for the ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery: a report of the International Brachial Artery Reactivity Task Force. J Am Coll Cardiol. 2002 Jan 16;39(2):257-65. doi: 10.1016/s0735-1097(01)01746-6. PMID 11788217
- [Background] Deng YB, Wang XF, Le GR, Zhang QP, Li CL, Zhang YG. Evaluation of endothelial function in hypertensive elderly patients by high-resolution ultrasonography. Clin Cardiol. 1999 Nov;22(11):705-10. doi: 10.1002/clc.4960221105. PMID 10554684